CLINICAL TRIAL: NCT00466856
Title: Clinical Trial of Sir-Spheres® in Patients With Symptomatic or Progressive Hepatic Metastases From Neuroendocrine Tumors
Brief Title: Internal Radiation Therapy in Treating Patients With Liver Metastases From Neuroendocrine Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: due to slow accrual
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Meranze, MD, Vice-Chair, Department of Radiology and Radiological Science; Professor of Radiology and Surgery; Interventional Radiologist, Vanderbilt-Ingram Cancer Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VICC GI 0365; VU-VICC-GI-0365
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: Head and Neck Cancer; Islet Cell Tumor; Metastatic Cancer; Pheochromocytoma
Keywords: neoplastic syndrome; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; thyroid gland medullary carcinoma; metastatic pheochromocytoma; recurrent islet cell carcinoma; liver metastases; recurrent pheochromocytoma; gastrinoma; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma
MeSH Terms: conditions — Head and Neck Neoplasms; Adenoma, Islet Cell; Neoplasm Metastasis; Pheochromocytoma; Neoplasms; Carcinoma, Medullary; Carcinoma, Islet Cell; Gastrinoma; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma | interventions — Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sir-Spheres (Experimental)
  Interventions: Drug: octreotide acetate; Radiation: yttrium Y 90 resin microspheres

INTERVENTIONS:
Drug: octreotide acetate — Lung/liver Ratio Dose of SIR-Spheres
  * <10% Administer full dose of SIR-Spheres
  * 10% to 15% Reduce dose of SIR-Spheres by 20%
  * 16% to 20% Reduce dose of SIR-Spheres by 40%
  * >20% Do not give SIR-Spheres
  Other Names: octreotide
Radiation: yttrium Y 90 resin microspheres — radiation
  Other Names: octreotide

SUMMARY:
RATIONALE: Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

PURPOSE: This phase II trial is studying how well internal radiation therapy works in treating patients with liver metastases from neuroendocrine tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine tumor response to selective internal radiation therapy with yttrium Y 90 resin microspheres (Sir-Spheres®) in patients with progressive liver metastases from neuroendocrine tumors.

Secondary

* Determine the toxicity of this treatment in these patients.
* Determine the symptomatic relief of patients treated with this regimen.
* Determine the health-related quality of life of patients receiving this treatment.

OUTLINE: Patients have an catheter placed into the hepatic artery percutaneously through the groin and then undergo selective internal radiation therapy with yttrium Y 90 resin microspheres (Sir-Spheres®) via the catheter on day 1. Patients also receive octreotide acetate IV 1 hour prior to, during, and 2 hours after Sir-Spheres® injection. Patients may undergo above treatment in another lobe of the liver (if each lobe is treated separately) 4 weeks later.

Patients undergo functional performance, health-related quality of life, and symptom severity assessment prior to initial treatment and after completion of study treatment.

After completion of study treatment, patients are followed periodically for at least 1 year.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically confirmed neuroendocrine tumor metastatic to the liver

  * Well-differentiated or moderately well-differentiated neuroendocrine tumors
* Measurable disease, defined as ≥ 1 unidimensionally measurable lesion ≥ 20 mm with conventional techniques or ≥ 10 mm with spiral CT scan
* Symptomatic disease, meeting one of the following criteria:

  * Refractory carcinoid symptoms, defined as Carcinoid Symptom Severity scale > 2 despite use of octreotide acetate at ≥ 200 mcg subcutaneously three times daily (or 20 mg intramuscularly once monthly) for ≥ 4 weeks
  * Evidence of radiographic progression with either of the following manifestations:

    * Moderate-severe right upper quadrant pain and unintentional weight loss > 10%
    * Decline in Karnofsky performance status > 10 points
* At least a 20% increase in the sum of the longest diameters of target lesions in the liver within the past 12 months
* No more than 75% replacement of normal liver by neuroendocrine tumor
* No more than 20% arteriovenous lung shunting on a technetium Tc 99m macro-aggregated albumin nuclear scan
* No equivocal, nonmeasurable, or nonevaluable liver metastasis

PATIENT CHARACTERISTICS:

* Karnofsky performance status 50-100%
* Life expectancy ≥ 6 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Creatinine ≤ 1.5 mg/dL
* Bilirubin ≤ 2.0 mg/dL
* Albumin ≥ 3.0 g/dL
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 65,000/mm³
* Hemoglobin > 9.0 g/dL
* INR ≤ 1.4
* No hepatic arterial anatomy that would preclude the administration of study treatment into the liver
* No nonmalignant disease that would preclude study participation
* No other malignancy within the past 5 years except for cured basal cell carcinoma of the skin or cured carcinoma in situ of the uterine cervix

PRIOR CONCURRENT THERAPY:

* Prior surgery, chemotherapy, or locally ablative technique for the liver cancer allowed
* No prior radiotherapy to the upper abdomen that includes the liver in the treatment field
* No investigational drug or agent/procedure (i.e., participation in another clinical trial) within the past 4 weeks
* No other specific anticancer treatment (other than octreotide acetate) during and for 3 months after completion of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2003-12; Primary Completion 2006-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Tumor response | at 1 year or until intervening death

SECONDARY OUTCOMES:
Toxicity as measured by CTC v3.0 | at 1 year or until intervening death
Symptomatic relief as measured by Carcinoid Symptom Scale, SF-36 Pain scale, and SF-36 physical component summary | at 1 year or until intervening death
  The Carcinoid Symptom Severity Scale is a self-report instrument that addresses the severity and frequency of symptoms and their impact on daily living.
Patient report of Health-related quality of life (HRQOL) | at 1 year or until intervening death
  HRQOL will be determined via the Medical Outcome Study 36-item short form, which includeds 8 individual scales, physical and mental component summary scores and is normed to both health and clinical populations.

CONTACTS AND LOCATIONS:
Overall Officials: Steven G. Meranze, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States